CLINICAL TRIAL: NCT04411030
Title: A Two Cohort, Open-Label, Fixed Sequence Study to Investigate the Effect of CYP3A4 Inhibition on the Single Dose Pharmacokinetics of ASTX660 and the Effect of a Single Dose of ASTX660 on the Pharmacokinetics of the CYP3A4 Substrate Midazolam
Brief Title: A Study to Investigate the Effect of CYP3A4 Inhibition on the Single Dose Pharmacokinetics of ASTX660 and the Effect of a Single Dose of ASTX660 on the Pharmacokinetics of the CYP3A4 Substrate Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: ASTX660-12
Record Dates: First submitted 2020-05-29; First posted 2020-06-01 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — ASTX-660; Midazolam; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Oral administration of ASTX660 and itraconazole at specific time points.
  Interventions: Drug: ASTX660; Drug: Itraconazole
- Part 2 (Experimental): Oral administration of ASTX660 and midazolam at specific time points.
  Interventions: Drug: ASTX660; Drug: Midazolam

INTERVENTIONS:
Drug: ASTX660 — Form: capsule; Route of administration: oral
Drug: Midazolam — Form: syrup; Route of administration: oral
  Arms: Part 2
Drug: Itraconazole — Form: capsule; Route of administration: oral
  Arms: Part 1

SUMMARY:
In Part 1, the primary objective is to investigate the effect of multiple doses of itraconazole, an inhibitor of CYP3A4, on the pharmacokinetic (PK) profile of a single dose of ASTX660.

In Part 2, the primary objective is to investigate the effect of a single dose of ASTX660 on the pharmacokinetics of the CYP3A4 substrate midazolam and its metabolite, 1-hydroxy midazolam.

Safety and tolerability of a single dose of ASTX660 in the absence and presence of multiple doses of the CYP3A4 inhibitor itraconazole and in the presence of a single dose of the CYP3A4 substrate midazolam will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Participant understands the study procedures and agrees to participate by providing written informed consent.
2. Participant is willing and able to comply with all study procedures and restrictions.
3. Participant is male aged 18 to 45 years, inclusive at Screening.
4. Participant has a body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 30.0 kg/m2 at Screening.
5. Participant is considered medically healthy as determined by the investigator, based on clinical evaluations including medical history, physical examination, clinical laboratory tests, 12-lead electrocardiogram (ECG) in triplicate, and vital sign measurements performed at Screening.
6. Participants must be willing to use adequate contraception (double-barrier) from screening until 3 months after study completion. Male vasectomy is accepted as contraception if the vasectomy took place ≥ 6 months prior to first dose.
7. Participants must refrain from sperm donation, from screening until 3 months after study completion.

Exclusion Criteria:

1. Participant is mentally or legally incapacitated or has significant emotional problems at the time of Screening or is expected to have such problems during the conduct of the study.
2. Participant has a clinically significant medical or psychiatric condition or disease (acute or chronic) that, as judged by the investigator, would make the participant ineligible for participation in the study (eg, compromises the study data, limits the participant's ability to complete and/or participate in the study).
3. Participant has a current condition or history of significant endocrine, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, immunological, or neurological disorders with clinical manifestations that, as judged by the investigator, would make the participant ineligible for participation in the study.
4. Participant has a chronic disease requiring medication, dietary restriction, physical therapy, and/or other routine treatment that, as judged by the investigator, would make the participant ineligible for participation in the study.
5. Participant has a history of gastrointestinal (GI) surgery including but not limited to gastric resection and/or intestinal resection that resulted in a clinically significant abnormality in GI function.
6. Participant has a history or presence of cancer (with the exception of a history of basal cell carcinoma of the skin).
7. Participant has a history of drug and/or alcohol addiction or is a current regular user (including recreational use) of any illicit drugs, has a history of drug or alcohol abuse, or has ever undergone drug or alcohol rehabilitation.
8. Participant has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerance to food, prescription drugs or non-prescription (over-the-counter) drugs. Note: participants with seasonal allergies may participate.
9. Participant has a known history of coronavirus disease 2019 (COVID-19) or has had contact with a severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positive or COVID-19 patient within the 4 weeks prior to admission to the study center.
10. Participant has a QTcF interval of > 450 msec at Screening.
11. Participant has an estimated creatinine clearance < 90 mL/min based on the Cockcroft Gault equation at Screening.
12. Participant regularly consumes excessive amounts of caffeine, defined as > 6 servings of coffee, tea, cola, or other caffeinated beverages, per day (1 serving is approximately equivalent to 120 mg of caffeine).
13. Participant regularly consumes excessive amounts of alcohol, defined as > 3 glasses of alcoholic beverages per day and/or refuses to refrain from consuming such products throughout the study.
14. Participant has used any medication (including prescription or non-prescription drugs, dietary or vitamin/mineral supplements or herbal remedies that are known to induce drug-metabolizing enzymes) within 14 days (or 5 half-lives, whichever is longer) prior to study drug administration on Day 1.
15. Participant has used any medications known to be significant CYP inducers, including St. John's wort, within 28 days prior to the study drug administration on Day 1.
16. Participant has consumed grapefruit, grapefruit juice, grapefruit juice-containing products, Seville oranges, orange juice, and/or apple juice within 7 days prior to study drug administration on Day 1 and/or refuses to refrain from consuming such products throughout the study.
17. Participant has consumed vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard) and/or charbroiled meats within 7 days prior to study drug administration on Day 1 and/or refuses to refrain from consuming such products throughout the study.
18. Participant has used tobacco- or nicotine-containing products (eg, cigarette, pipe, cigar, chewing, nicotine patch, or nicotine gum) within 6 months prior to Day -1.
19. Participant refuses to refrain from using tobacco- or nicotine-containing products throughout the study.
20. Participant has a positive urine drug and/or alcohol screening test result at Screening or on Day -1.
21. Participant has a positive test result for any serological test including human immunodeficiency virus (HIV) antigen/antibody, Hepatitis B surface antigen (HBsAg), and Hepatitis C virus (HCV) antibody at Screening.
22. Participant has a positive test result for SARS-CoV-2 antigen, either asymptomatic or present with COVID-19 at study check-in.
23. Participant appears to have poor venous access.
24. Participant has donated blood or had significant blood loss within 56 days of study drug administration on Day 1.
25. Participant has donated plasma within 7 days prior to study drug administration on Day 1.
26. Participant has participated in any other investigational trial or has received any investigational drug within 28 days (or 5 half-lives of the previous investigational drug). The date will be derived from the last study procedure [blood collection or dosing] of previous trial prior to study drug administration on Day 1.
27. Participant has any hypersensitivity to the study drugs or any of their excipients.
28. Participant is ineligible for this study for any other reason, as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of ASTX660: Cmax | From predose up to Day 14
  Maximum plasma concentration
Pharmacokinetic parameter of ASTX660: AUC0-t | From predose up to Day 14
  Area under the plasma concentration versus time curve from time zero to the last measurable concentration
Pharmacokinetic parameter of ASTX660: AUC0-24 | From predose up to Day 14
  Area under the plasma concentration versus time curve from time zero to 24 hours
Pharmacokinetic parameter of ASTX660: AUC0-inf | From predose up to Day 14
  Area under the plasma concentration versus time curve from time zero extrapolated to infinity
Pharmacokinetic parameter of midazolam and 1-hydroxyl midazolam: Cmax | From predose up to Day 9
  Maximum plasma concentration
Pharmacokinetic parameter of midazolam and 1-hydroxyl midazolam: AUC0-t | From predose up to Day 9
  Area under the plasma concentration versus time curve from time zero to the last measurable concentration
Pharmacokinetic parameter of midazolam and 1-hydroxyl midazolam: AUC0-24 | From predose up to Day 9
  Area under the plasma concentration versus time curve from time zero to 24 hours
Pharmacokinetic parameter of midazolam and 1-hydroxyl midazolam: AUC0-inf | From predose up to Day 9
  Area under the plasma concentration versus time curve from time zero extrapolated to infinity

SECONDARY OUTCOMES:
Pharmacokinetic parameter for ASTX660: CL/F | From predose up to Day 14
  Total apparent clearance
Pharmacokinetic parameter for ASTX660: t1/2 | From predose up to Day 14
  Observed terminal half-life
Pharmacokinetic parameter for midazolam: CL/F | From predose up to Day 9
  Total apparent clearance
Pharmacokinetic parameter for midazolam: t1/2 | From predose up to Day 9
  Observed terminal half-life
Safety: Number of participants with adverse events | Up to Day 35

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Bio-kinetic, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No